CLINICAL TRIAL: NCT01810458
Title: Clinical Predictors and Epigenetic Markers for Liver Fibrosis in Alpha-1 Antitrypsin Deficiency
Brief Title: Liver Fibrosis in Alpha-1 Antitrypsin Deficiency (Liver AATD)
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201601019; 910 (Other: Clinical Research Center at Shands UF); IRB201601019/ 63-2013 (Other: Univeristy of Florida)
Record Dates: First submitted 2013-03-06; First posted 2013-03-13 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Liver Fibrosis; Alpha-1 Antitrypsin Deficiency; AAT Deficiency; AATD
Keywords: Liver; Fibrosis; Alpha-1; AAT; AATD
MeSH Terms: conditions — Liver Cirrhosis; alpha 1-Antitrypsin Deficiency; Fibrosis | interventions — Health Records, Personal; Restraint, Physical; Blood Specimen Collection; Phlebotomy; Surveys and Questionnaires; Biopsy; Midazolam; Fentanyl; Lidocaine; Acetaminophen; Lorazepam; oxycodone-acetaminophen; Ondansetron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver tissue and whole blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AATD ZZ and Rare Alleles Group: Participants will get a history and physical (H&P) and have an intravenous catheter (IV) placed, for blood draws, at the screening and years 1-3 visits. An IV will also be placed at the liver biopsy visit(s) for the administration of medication. An abdominal ultrasound will be done at the screening and year 3 visits along with the completion of a liver questionnaire. Finally, participants will have a liver biopsy done, with the use of lidocaine, lorazepam, or midazolam and fentanyl, after the screening visit and potentially at the year 3 study visit, depending on the results of the first liver biopsy. Participants who experience pain after the liver biopsy may receive acetaminophen or oxycodone/acetaminophen. Any subject experiencing nausea may receive ondansetron.
  Interventions: Device: Abdominal ultrasound; Procedure: History and physical; Procedure: Intravenous catheter; Procedure: Blood draw; Other: Liver questionnaire; Procedure: Liver Biopsy; Drug: Midazolam; Drug: Fentanyl; Drug: Lidocaine; Drug: Acetaminophen; Drug: Lorazepam; Drug: Oxycodone/Acetaminophen; Drug: Ondansetron

INTERVENTIONS:
Device: Abdominal ultrasound — Abdominal ultrasound will be done at the liver biopsy visits. The purpose of the ultrasound is to evaluate for the presence of liver fibrosis and identify the biopsy site.
  Other Names: SonoSite Edge Ultrasound System
Procedure: History and physical — Every study participant will be asked about their medical history and will have a physical exam done at the screening, year 1, year 2, and year 3 visits.
  Other Names: H&P; exam; medical history
Procedure: Intravenous catheter — Every study participant will have and intravenous catheter (IV) placed at every study visit. The IV will be used for the collection of blood at the screening, year 2, year 2, and year 3 visits. It will also be used for the administration of medication at the first liver biopsy, as well as the year 3 visit if the biopsy is repeated.
  Other Names: IV
Procedure: Blood draw — At the screening, year 1, year 2, and year 3 visits, every participant will have blood collected from the IV that is placed in one of their veins.
  Other Names: Phlebotomy
Other: Liver questionnaire — At the screening and year 3 visits, every subject will complete a questionnaire which involves questions regarding liver health.
  Other Names: Questionnaire
Procedure: Liver Biopsy — Every participating subject who passes the screening visit, will have a liver biopsy done with the use of lidocaine (a numbing medicine) injected into skin where the biopsy will be collected. At the time of the biopsy, either lorazepam (a medicine used to treat anxiety and cause relaxation) or midazolam (a medicine used to cause sleepiness and amnesia) and fentanyl (a medicine used to relieve pain) will be used. Once the relaxation medication and numbing medicine have been given, a sample of liver tissue will be collected using a needle biopsy device.
  Other Names: Biopsy
Drug: Midazolam — Every participating subject who passes the screening visit, will have a liver biopsy done with the use of lidocaine injected into skin where the biopsy will be collected. At the time of the biopsy, either lorazepam (a medicine used to treat anxiety and cause relaxation) or midazolam (a medicine used to cause sleepiness and amnesia) and fentanyl (a medicine used to relieve pain) will be used. After the biopsy is done, participants who continue to have pain may receive either oxycodone/acetaminophen or acetaminophen (medicines used to relieve pain). Any participant who experiences nausea may receive ondansetron (a medicine used to relieve nausea).
  Other Names: Versed
Drug: Fentanyl — Every participating subject who passes the screening visit, will have a liver biopsy done with the use of lidocaine injected into skin where the biopsy will be collected. At the time of the biopsy, either lorazepam (a medicine used to treat anxiety and cause relaxation) or midazolam (a medicine used to cause sleepiness and amnesia) and fentanyl (a medicine used to relieve pain) will be used. After the biopsy is done, participants who continue to have pain may receive either oxycodone/acetaminophen or acetaminophen (medicines used to relieve pain). Any participant who experiences nausea may receive ondansetron (a medicine used to relieve nausea).
  Other Names: Fentora; Onsolis
Drug: Lidocaine — Every participating subject who passes the screening visit, will have a liver biopsy done with the use of lidocaine injected into skin where the biopsy will be collected. At the time of the biopsy, either lorazepam (a medicine used to treat anxiety and cause relaxation) or midazolam (a medicine used to cause sleepiness and amnesia) and fentanyl (a medicine used to relieve pain) will be used. After the biopsy is done, participants who continue to have pain may receive either oxycodone/acetaminophen or acetaminophen (medicines used to relieve pain). Any participant who experiences nausea may receive ondansetron (a medicine used to relieve nausea).
  Other Names: Xylocaine
Drug: Acetaminophen — Every participating subject who passes the screening visit, will have a liver biopsy done with the use of lidocaine injected into skin where the biopsy will be collected. At the time of the biopsy, either lorazepam (a medicine used to treat anxiety and cause relaxation) or midazolam (a medicine used to cause sleepiness and amnesia) and fentanyl (a medicine used to relieve pain) will be used. After the biopsy is done, participants who continue to have pain may receive either oxycodone/acetaminophen or acetaminophen (medicines used to relieve pain). Any participant who experiences nausea may receive ondansetron (a medicine used to relieve nausea).
  Other Names: Tylenol
Drug: Lorazepam — Every participating subject who passes the screening visit, will have a liver biopsy done with the use of lidocaine injected into skin where the biopsy will be collected. At the time of the biopsy, either lorazepam (a medicine used to treat anxiety and cause relaxation) or midazolam (a medicine used to cause sleepiness and amnesia) and fentanyl (a medicine used to relieve pain) will be used. After the biopsy is done, participants who continue to have pain may receive either oxycodone/acetaminophen or acetaminophen (medicines used to relieve pain). Any participant who experiences nausea may receive ondansetron (a medicine used to relieve nausea).
  Other Names: Ativan
Drug: Oxycodone/Acetaminophen — Every participating subject who passes the screening visit, will have a liver biopsy done with the use of lidocaine injected into skin where the biopsy will be collected. At the time of the biopsy, either lorazepam (a medicine used to treat anxiety and cause relaxation) or midazolam (a medicine used to cause sleepiness and amnesia) and fentanyl (a medicine used to relieve pain) will be used. After the biopsy is done, participants who continue to have pain may receive either oxycodone/acetaminophen or acetaminophen (medicines used to relieve pain). Any participant who experiences nausea may receive ondansetron (a medicine used to relieve nausea).
  Other Names: Percocet; Tylox
Drug: Ondansetron — Every participating subject who passes the screening visit, will have a liver biopsy done with the use of lidocaine injected into skin where the biopsy will be collected. At the time of the biopsy, either lorazepam (a medicine used to treat anxiety and cause relaxation) or midazolam (a medicine used to cause sleepiness and amnesia) and fentanyl (a medicine used to relieve pain) will be used. After the biopsy is done, participants who continue to have pain may receive either oxycodone/acetaminophen or acetaminophen (medicines used to relieve pain). Any participant who experiences nausea may receive ondansetron (a medicine used to relieve nausea).
  Other Names: Zofran

SUMMARY:
We hypothesize that individuals with Alpha-1 Antitrypsin (AAT) deficiency have ongoing liver injury which is not detected by the usual blood tests used to look at liver function. This ongoing liver injury leads to cirrhosis in a significant number of adults with AAT deficiency.

DETAILED DESCRIPTION:
Our overarching hypothesis is that liver disease in adults with AAT deficiency is the result of the accumulation of the abnormally folded protein within the endoplasmic reticulum of the hepatocyte. In some individuals, the intrinsic cellular mechanisms of the hepatocyte are sufficient to clear adequate amounts of the abnormally folded protein such that liver disease does not occur. In AAT deficient individuals who develop liver disease, environmental and other genetic factors stress the hepatocyte, and the normal cellular mechanisms that maintain homeostasis are disrupted, leading to liver disease.

For this proposal, our hypothesis is that the prevalence of liver disease in adults with AAT is higher than previously reported because liver injury and fibrosis is not accurately detected by available routine liver testing. Testing this hypothesis will require an initial evaluation for liver disease with liver function testing and imaging, and then histologic confirmation by liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Alpha-1 Antitrypsin deficiency confirmed to be PI*ZZ by both genotype or another identified rare allele;
* Age range from 18-70;
* Willingness to consent to liver biopsy;
* Ability to travel to UF as necessary by protocol; and
* Platelet count greater than or equal to 50,000/mm3 and an INR less than or equal to 1.5.

Exclusion Criteria:

* Hemophilia, anticoagulant therapy that cannot be interrupted briefly, malignancy, or any other condition that would compromise the safety of a liver biopsy;
* Any known pre-existing medical condition that might interfere with the patient's participation in and completion of the study or any condition, which in the opinion of the investigator would make the patient unsuitable for enrollment;
* Active substance abuse including, but not limited to, alcohol, intravenous or, inhaled drugs;
* History of adverse reactions or allergy to the local anesthetic, sedative, or pre-medication used for the percutaneous liver biopsy;
* Poor venous access making the subject unable to complete the required laboratory testing schedule; and
* Females who are pregnant or lactating at time of enrollment. Should a female subject become pregnant during the follow up period after the initial liver biopsy, continued participation would be allowed if the following conditions are met: the subject desires to continue; a discussion of risk and benefits of participation between the principal investigator and the subject has occurred; and no liver biopsy would be performed in the follow up period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonary clinic, hepatology clinic, and the Alpha-1 Antitrypsin Tissue and Data Bank.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
To estimate the prevalence and histologic spectrum of liver injury in an adult with Alpha-1 Antitrypsin deficiency having a ZZ genotype or other rare allele. | up to 30 days
  An abdominal ultrasound will be done at the screening visit. A liver biopsy will be done on subjects who pass the screening process. The biopsy will be done within 30 days of the screening visit.

SECONDARY OUTCOMES:
To identify environmental and host risk factors for clinically significant liver fibrosis. | At each study visit including screening, first liver biopsy, year 1, year 2, and year 3 visits.
  A liver disease questionnaire will be done at the time of the first liver biopsy and at the year 3 study visit. A history and physical will also be completed at the screening visit, year 1 visit, year 2 visit, and year 3 visit.
To define the diagnostic accuracy of non-invasive markers of fibrosis in AAT liver disease. | At the screening and year 3 visits.
  An abdominal ultrasound will be completed at the screening visit and the year 3 visit.
To explore epigenetic markers for the development of liver fibrosis. | Starting with the first liver biopsy and ending with the second liver biopsy done at year 3.
  Liver tissue collected at the time of the first biopsy will be sent for testing which will evaluate for epigenetic markers of liver fibrosis. For subjects whose initial liver biopsy reveals liver fibrosis between stages 2 - 4, additional liver tissue will be collected at the time of the repeat biopsy done at the year 3 study visit.
To quantify liver fibrosis progression. | At each study visit including screening, first liver biopsy, year 1, year 2, and year 3 visits.
  The presence and progression of liver fibrosis will be evaluated by an abdominal ultrasound done at the screening visit, year 1 visit, year 2 visit, and year 3 visit. A liver biopsy will be done if a subject passes the screening visit and will be repeated at the year 3 study visit if the initial liver biopsy reveals liver fibrosis between stages 2 - 4.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Brantly, MD, Principal Investigator — University of Florida
Locations (1):
- Shands at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Enrolled subjects will receive copies of all their clinical testing done while enrolled in the study. Otherwise, all data for publication purposes will be de-identified.

REFERENCES:
- [Derived] Clark VC, Marek G, Liu C, Collinsworth A, Shuster J, Kurtz T, Nolte J, Brantly M. Clinical and histologic features of adults with alpha-1 antitrypsin deficiency in a non-cirrhotic cohort. J Hepatol. 2018 Dec;69(6):1357-1364. doi: 10.1016/j.jhep.2018.08.005. Epub 2018 Aug 21. PMID 30138687